CLINICAL TRIAL: NCT02635022
Title: Fragility Fracture Liaison Service and Anti-osteoporosis Medication Monitoring Service Study in Rural Area
Brief Title: Fragility Fracture Liaison Service and Anti-osteoporosis Medication Monitoring Service Study
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201506039RIND
Record Dates: First submitted 2015-11-25; First posted 2015-12-18 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis; Fracture
Keywords: Fracture; Sarcopenia; Osteoporosis; Care management; Medication adherence
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; Sarcopenia; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FLS: Patients with new hip fracture or newly identified vertebral fractures
- MMS: Patients prescribed with anti-osteoporosis medications but not fit FLS requirements

SUMMARY:
Aims: (1) to Establish the FLS services at the National Taiwan University Hospital Jinshan Branch. (2) To establish a anti-osteoporosis medication management service at Jinshan Branch.

Method: From Aug., 2015, a fracture liaison services (FLSs) following the 13 'Capture the Fracture Best Practice Standards' were implemented at the National Taiwan University Hospital Jinshan Branch health care system. The Jinshan Branch program enrolled patient with 1) new hip fracture 2) newly identified vertebral fractures (radiological or clinical) from both inpatients and outpatients. At the same time, a osteoporosis medication management service is also establish as a complement of FLS to enroll patients on antiosteoporosis medications (AOMs) but not necessary with fracture.

Participating physicians will select those eligible for services and refer to study coordinators. Study coordinators will conduct baseline assessments on osteoporosis/fracture risks, record medical conditions, AOMs, provide educations on osteoporosis, fracture, sarcopenia, fall, medications, nutrition, and exercise. They also arrange return clinic visit, telephone reminder and follow up for patients, and communicate with providers on regular bases.

During the whole study period, the investigators planed to enroll 200 patients (with or without fracture). Each patient would be assessed at baseline, and every 4 months last for two years.

DETAILED DESCRIPTION:
Background:The Asia Fracture Gap Taiwan Study (AFGTS) showed that among fragility fracture sufferers, only 1/4 of them underwent bone mineral density (BMD) tests and 1/3 of them received treatments for osteoporosis. Secondary fragility fracture prevention services are needed to improve the care gaps. In addition, one-year adherence to oral anti-osteoporosis medication (AOMs) was only about 30%. In recent years, efforts have been made to change the delivery of these medications from oral form to injection form every, 3, 6 or 12 months to increase adherence. However, both patients and providers are sometimes confused about the multiple choices. Also, patients may receive extra medications if providers did not keep tract of their previous AOM uses or patients may changes providers. There were urgent needs to provide AOM monitoring and management services to improve cares.

. Aims: (1) to Establish the FLS services at the National Taiwan University Hospital Jinshan Branch. (2) To establish a anti-osteoporosis medication management service at Jinshan Branch.

Method: The FMS was designed following the 13 'Capture the Fracture Best Practice Standards'. The National Taiwan University Hospital (NTUH) institutional review board approved the study in Aug., 2015. Patients were eligible to be enrolled into the FMS part of the study if they had

* Age >=50 and one of the below
* New hip fracture in orthopedic ward
* Newly identified radiographic vertebral fractures from plan films in geriatric ward or clinical vertebral fractures in outpatient clinics
* Newly prescribed with AOMs
* Recent change of AOMs
* Poor adherence to AOMs
* Participating physicians feel that the service will benefit the patient in overall osteoporosis and medication managements.

Exclusion Criteria:

* Life expectancy less than 2 years or can't be assessed for communication problems
* Atypical fractures
* Patient in other medication clinical trials
* Unwilling to accept the assessment and treatment

Osteoporosis-related assessments, treatments, consultations on diet, medications, exercise, fall prevention were given mainly by care managers. A system is set up to remind patients to take their medications at home or to return to clinic for regular injections of medications. Follow up assessments included adherence to education instructions, medications, fall and fracture incidences. During the whole study period, we planed to enroll 200 patients. Each patient would be assessed at baseline, and every 4 months last for two years.

Anticipated results:

Establish Osteoporosis-related patient database combined with NTUH Participating physicians and care managers will learn new skills in managing osteoporosis patients.

Enhance adherence to AOMs The results published in the International Osteoporosis Conferences

ELIGIBILITY:
Inclusion Criteria:

* Age >=50 and one of the below
* New hip fracture in orthopedic ward
* Newly identified radiographic vertebral fractures from plan films in geriatric ward or clinical vertebral fractures in outpatient clinics
* Newly prescribed with AOMs
* Recent change of AOMs
* Poor adherence to AOMs
* Participating physicians feel that the service will benefit the patient in overall osteoporosis and medication managements.

Exclusion Criteria:

* Life expectancy less than 2 years or can't be assessed for communication problems
* Atypical fractures
* Patient in other medication clinical trials
* Unwilling to accept the assessment and treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: new fragility fracture Adults treated with anti-osteoporosis medicines (AOMs)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes of medication adherence | 12 MONTHS
  Changes of medication adherence for all participants will be assessed at the 4, 8, 12, 18 and 24 months after enrollments. However, the main primary outcome will be set at the adherence at 12 months. If the patient changes medication, all AOMs adherence will be combined.
  Specific formulas of medication adherence assessments are as below:
  1. for oral medications: adherence is defined as: medication taken/ medication prescribed within past 3 months
  2. for injection medications: adherence is defined as: of injection/ of due injection since baseline or last follow up phone call. Statistics: Simple counts of adherence (%) among all participants.

SECONDARY OUTCOMES:
The proportion of patients received Bone Mineral Density test within 8 week after enrollments | 8 week
  This outcome is concerned with the percentage of FLS patients received BMD test at the timing (8 week) of when post-fracture assessment is done.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital, Chutung branch
Locations (1):
- National Taiwan University Hospital, Chutung branch, Hsinchu, Taiwan